CLINICAL TRIAL: NCT02171325
Title: A Phase Ⅱ Study of Different Doses of Irinotecan and Cisplatin for First-line Extensive-stage Small-cell Lung Cancer Treatment
Brief Title: Study of Different Doses of Irinotecan and Cisplatin for First-line Extensive-stage Small-cell Lung Cancer Treatment
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guangdong Association of Clinical Trials (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTONG1402
Record Dates: First submitted 2014-06-16; First posted 2014-06-24 (Estimated); Last update posted 2021-02-03 (Actual); Status verified 2021-02

CONDITIONS: Small Cell Lung Cancer
Keywords: irinotecan; Small Cell Lung Cancer
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- irinotecan (Experimental): irinotecan； 60 mg/m2、65mg/m2、70mg/m2、75mg/m2、80mg/m2、85mg/m2、90mg/m2、95mg/m2、100mg/m2
  Interventions: Drug: irinotecan

INTERVENTIONS:
Drug: irinotecan — 60 mg/m2、65mg/m2、70mg/m2、75mg/m2、80mg/m2、85mg/m2、90mg/m2、95mg/m2、100mg/m2

SUMMARY:
The purpose of this study is to identify the appropriate dose of irinotecan by dose escalation(dose climbing) test. The study would provide rationale for regimen decision in a future phase III clinical trial, in which irinotecan combined with cisplatin(IP) will be selected as therapeutic drugs.

DETAILED DESCRIPTION:
To determine the Maximum Tolerated Dose (MTD) and Limiting Toxicity (DLTs) of irinotecan in patients with extensive stage small cell lung cancer treated with irinotecan plus cisplatin

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 to 65 years, male and female
2. Histologically or cytologically confirmed extensive stage .small cell lung cancer(SCLC )（except metastases only as pleural effusion）
3. No prior chemotherapy
4. Metastatic lesion had been treated more than 14 days by palliative radiation therapy or surgery
5. With measurable tumor lesions (Non-irradiated parts),(RECIST 1.1: Without radiotherapy ,the longest diameter is more than 10mm by CT or MRI ,except that lymph nodes need short diameter need more then 15mm, and the lesions can be accurately evaluated repeatedly measurable)
6. Eastern Cooperative Oncology Group(ECOG) Performance Status 0-1
7. Expected survival ≥ 3months
8. Marrow,kidney, liver,heart and lung are well -functioning,and absolute count of

   * absolute neutrophil coun(ANC) ≥ 2.0 × 109 / L
   * blood platelet(PLT) ≥ 100 × 109 / L
   * Hb≥ 90g / L
   * conjugative bilirubin(CB)≤ upper limit of normal(ULN) × 1.5
   * Aspartate transaminase(AST )(glutamic oxalacetic transaminase,GOT): ≤ upper limit of normal(ULN )× 2.5
   * Alanine aminotransferase(ALT)(Glutamate Pyruvate Transaminase,GPT): ≤ ULN × 2.5
   * Serum creatinine: ≤ ULN or calculated creatinine clearance≥ 60 ml / min
   * (PT INR) ≤ ULN × 1.5
   * ECG: no abnormalities in need of treatment
9. No pregnancy or no pregnancy demand at the end of the study within six months
10. Must provide written informed consent.

Exclusion Criteria:

1. Patient have platinum compounds allergy history
2. Patient with active ulcer disease or chronic enteritis patients
3. Primary lesion(s) has (have) been treated by Surgery or radiation
4. Patient had received Immune drugs treatment for anti-lung cancer indications or anti-cancer Chinese traditional medicine treatment within two weeks
5. Patients with interstitial pneumonia or pulmonary fibrosis
6. Brain metastasis requiring treatment
7. Patient with bronchus or bronchial stenosis or blockage and superior vena cava syndrome caused by serious invasion
8. Patients with severe infections, severe abnormal secretion of (Anti Diuretic Hormone,ADH) syndrome, poorly controlled diabetes, severe complications requiring treatment vena cava syndrome
9. Severe cardiovascular disease: hypertension that medical treatment can not be controlled , unstable angina, myocardial infarction within the last June a history of congestive heart failure> 3 (NYHA) and severe arrhythmia

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2014-06; Primary Completion 2021-06 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Limiting Toxicity (DLT )in the irinotecan | up to 18 weeks

SECONDARY OUTCOMES:
Maximum Tolerated Dose(MTD)in the irinotecan | up to 18weeks

CONTACTS AND LOCATIONS:
Overall Officials: ying cheng, doctor, Principal Investigator — Jilin Provincial Tumor Hospital
Locations (1):
- Jilin cancer hospital, Changchun, Jilin, China

IPD SHARING:
Plan to Share IPD: No